CLINICAL TRIAL: NCT05708547
Title: Role of Mitophagy in Myeloid Cells During Coronary Atherosclerosis.
Acronym: MITOCARDIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NUGUYEN AOI 2022
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atheromatous coronary patients: patients scheduled for coronary artery bypass surgery with extracorporeal circulation
  Interventions: Biological: Blood samples; Procedure: myocardial tissue samples; Other: Data collection
- Non-atheratomous patients: Patients scheduled for valve or ascending aorta surgery with extracorporeal circulation without coronary lesion or peripheral arterial disease
  Interventions: Biological: Blood samples; Procedure: myocardial tissue samples; Other: Data collection

INTERVENTIONS:
Biological: Blood samples — at the beginning of the extracorporeal circulation, at the end of the extracorporeal circulation and at D1
Procedure: myocardial tissue samples — use of usually harvested right auricular tissue
Other: Data collection — pre-operative data: demographic data, severity scores, co-morbidities, treatments administered, collection of the presence and stage of arteriosclerotic disease, SYNTAX score Collection of data on the procedure Data from the clinical evaluation and daily biological examinations until D7 data from the follow-up consultation between D30 and D60: late complications, total length of stay in intensive care and hospital

SUMMARY:
Atherosclerosis (deposition of a plaque essentially composed of lipids on the artery walls) is a frequent condition and is a leading cause of death worldwide. In addition to the long-established risk factors such as age, hypertension, diabetes or sedentary lifestyle, it has been demonstrated that immune cells can participate in the genesis of atherosclerotic plaques through metabolic and mitochondrial reprogramming.

A non-invasive marker of this immune reprogramming has yet to be identified. Through the comparison of a group of atheromatous patients and a group of non-atheromatous patients, this study aims to evaluate this reprogramming phenomenon using a novel non-invasive method.

This monocentric interventional study will take place at the Dijon Bourgogne University Hospital and will include 50 patients divided into 2 groups: "atheromatous coronary patients" and "non-atheromatous patients". The duration of participation in this study is 1 month. This study is based on usually performed procedures. Only blood samples will be taken on a catheter usually used during any cardiac surgery in addition to the medical care that is provided during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

- Person who provides oral consent

Group 1:

- Patient scheduled for cardiac bypass surgery (isolated procedure) with extracorporeal circulation

Group 2:

* Patient scheduled for valve ou ascending aorta surgery with extracorporeal circulation
* No coronary lesion
* No peripheral arterial disease (limbs, carotids, aortic aneurysm)

Exclusion Criteria:

* Person not affiliated with national health care system
* Medication that alters mitochondrial function (Chloroquine, hydroxychloroquine, rapamycin, carbamazepine, resveratrol, sildenafil)
* Person under a legal protection measure (curatorship, guardianship, tutorship)
* Pregnant, parturient or breastfeeding women
* Major unable to express consent
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atheromatous coronary patients and non-coronary patients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Mitophagy level by flow cytometry | Before the introduction of extracorporeal circulation.
  Average fluorescence corresponding to PINK1-AF488 intracellular labelling (mitophagy checkpoint) in conventional (CD33+, CD66b-, CD14++, CD16-), intermediate (CD33+, CD66-, CD14++, CD16+), or non-conventional (CD33+, CD66b-, CD14+, CD16++) monocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France